CLINICAL TRIAL: NCT02023073
Title: Study of Physical Parameters Related to Laser Radiation and Its Interaction With Different Parts of the Human Eye
Brief Title: Determination of Physical Parameters Relevant to Ophthalmic Lasers
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ygal Rotenstreich, Director, Electrophysiology Clinic, Goldschleger Eye Research Institute, Sheba Medical Center
Other Study IDs: SHEBA-13-9977-YR-CTIL
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers

SUMMARY:
The use of lasers in medicine in general, and diagnosis and treatment in ophthalmology in particular, increased significantly. Making retinal surgery using lasers have become increasingly common. The goal: to diagnose eye diseases safely

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Refraction up to ±0.25D,
* General good health
* Written informed consent to participate in the study.

Exclusion Criteria:

* known current ophthalmic pathology
* known past ophthalmic pathology (including LASIK surgery)
* eye glasses or contact lenses

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Reflected laser radiation (Watt/cm 2) | 1 day
  The amplitude of laser radiation reflected from the eye at different wavelengths (532nm, 800nm & 900nm) at 4 angles (-10, 05, 0 and 10 degrees ) will be measured (Watt/cm 2)

SECONDARY OUTCOMES:
Reflection of laser radiation from the cornea (Watt/cm2) | 1 day
Reflection of laser radiation from the retina (Watt/cm 2) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ygal Rotenstreich, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Goldschleger Eye Research Institute, Sheba Medical Center,, Tel Litwinsky, Israel